CLINICAL TRIAL: NCT03627949
Title: The Effectiveness of an E-Intervention on Health Behavior Promotion in Chinese University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Yanping DUAN, Assistant Professor, Dr. Duan, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRG2/15-16/032
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Health Behavior; Physical Activity; Healthy Diet
Keywords: Web-based intervention; Health behavior change; University students; Health Action Process Approach Model
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Students in the intervention group 1 received first 4-week treatment on physical activity followed by 4-week treatment on healthy dietary behaviour.
  Interventions: Behavioral: E-intervention
- Intervention group 2 (Experimental): Students in the intervention group 2 received first 4-week treatment on healthy dietary behaviour followed by 4-week treatment on physical activity.
  Interventions: Behavioral: E-intervention
- Control group (No Intervention): Students in the control group were not provided with any supportive treatments on physical activity or healthy dietary behaviour.

INTERVENTIONS:
Behavioral: E-intervention — The intervention will address the basic elements of the HAPA model via the use of behaviour change techniques. In line with Abraham and Michie (2008), we use several behaviour change techniques like providing information about behavioural risk and benefit of behaviour change, prompting intention formation, prompting barrier identification, providing instructions how to perform a behaviour, prompting specific goal setting and review of behavioural goals, providing feedback on performance, prompting practice and providing follow-up prompts, prompting to plan social support and finally prompting relapse prevention, also based on strategies used by other effective computer tailoring programs. Students attended e-health intervention session once a week with about 20 minutes each time.
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
Through the internet and mobile phone SMS technology, and by using the Health Action Process Approach model as a theoretical backdrop, this 8-week theory-based intervention study aimed at developing a healthy lifestyle by supporting physical activity (PA) and a healthy dietary for Chinese university students. The investigators would examine whether the two intervention groups improve the participants' motivation for PA and healthy diets in comparison to the control group; whether, with the help of an intervention program, students are able to increase the PA levels and healthy diet consumption, and whether there are different effects between the two intervention programs.

DETAILED DESCRIPTION:
For the main study, the sample size was estimated by using G*Power 3.1 software with MANOVA approach (repeated measure). For achieving small effect size of 0.15 (Lippke, Fleig, Wiedemann, & Schwarzer, 2015), with a power (1-β) of 0.8 and alpha of 0.05, the total sample size was 306. Assuming a drop-out rate of approximately 30%, a total of 399 participants were required for the study evaluation.

The effects of the intervention were evaluated by performing several analyses of MANOVA and MANCOVA measured at three points in time (8-week apart pre-post measures, and four weeks follow-up; T1-T3).In addition, moderated multiple mediation analysis was performed (Independent variable: intervention; Moderators: stage; Dependent variable: behavioural and social-cognitive outcomes). Baseline characteristics of participants who dropped out were compared with participants who finished the intervention to examine whether drop out is at random or determined by specific characteristics.

ELIGIBILITY:
Inclusion Criteria:

* not professional athletes; not vegetarians
* no contraindication with respect to the physical activity or fruit and vegetable consumption.
* access to the Internet and a mobile phone.

Exclusion Criteria:

* have the restriction of physical mobility
* have fruit-vegetable related diseases such as diabetes or fruit allergies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change of weekly amount of physical activity (PA) | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  The level of PA will be measured through the short Chinese version of the IPAQ questionnaire (Macfarlane et al., 2007). Participants will be asked to estimate the number of days and hours spent for vigorous, moderate and walking activities during the past week.
Change of daily portions of fruit-vegetable intake (FVI) | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  The daily portions of FVI will be measured with four items, including fruit or vegetable juice, fruit, cooked or steamed vegetables, and raw vegetables (Rafferty et al., 2002). Respondents will be asked to count the number of portions of fruit and vegetables they consumed on average during a typical day.

SECONDARY OUTCOMES:
Change of stage algorithm of behaviors change | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  For PA, participants will be asked "Please think about your typical weeks: Did you engage in PA at least 5 days per week for 30 minutes or more?" Regarding dietary, participants will be asked "Please think about what you have typically consumed during the last weeks: Did you eat five portions of fruit and vegetables per day?" Responses are based on a rating scale with verbal anchors ("No, and I do not intend to start"; "No, but I am considering it"; "No, but I seriously intend to start"; "Yes, but only for a brief period of time"; "Yes, and for a long period of time") and are designed like a rating scale (Lippke, Ziegelmann, Schwarzer, & Velicer, 2009).
Change of outcome expectancies of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Outcome expectancies will be measured by two Pros items and two Cons items for each behavior (Schwarzer, Lippke, & Luszczynska, 2011).
Change of self-efficacy of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Self-efficacy will be assessed with three dimensions consisting of motivational, maintenance and recovery self-efficacies with the stem "I am certain that…" followed by 5 items for PA such as "…I can be physically active permanently at a minimum of 5 days a week for 30 minutes even if it is difficult", or followed by 5 items for FVI such as "…I can eat 5 portions of fruit and vegetable a day even if it is difficult." (Luszczynska & Sutton, 2006).
Change of risk perception of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Risk perception is adapted from Perloff and Fetzer (1986) and will be measured by 5 items.
Change of intention of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Intention will be assessed by 3 items for each behavior (Lippke et al., 2009).
Change of planning of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Planning will be distinguished into action planning and coping planning. Action planning will be assessed by 3 items for each behavior. Coping planning will be assessed by 3 items for each behavior (Schwarzer, 2008)
Change of perceived social support of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  For the perceived social support, the scale will be measured with the stem as "How do you perceived your environment?" followed by 3 items for PA such as"….People like my friends help me to stay physically active", or followed by 3 items for FVI such as "…People like my friends help me to eat healthily" (Jackson, Lippke & Gray, 2011).
Change of compensatory health beliefs of PA and FVI | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  Compensatory health beliefs will be measured by 4 items (Knäuper, Rabiau, Cohen, & Patriciu, 2004).
Change of perceived quality of life | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  This indicator will be assessed by using the short version of WHO Quality of Life-BREF (WHO, 1993). Respondents will be firstly asked about their general quality of life as "How would you rate your quality of life?", then 7 items in physical health sub-domain will be used, such as the example item "To what extent do you feel that physical pain prevents you from doing what you need to do?"
Change of body mass index (BMI) | From baseline to 9 weeks (at the end of intervention) and 1-month follow-up
  The participants will be asked to report body height (in cm) and body weight (in kg) for calculate the BMI.

OTHER OUTCOMES:
Demographic information | At baseline
  These items include gender, age, study year, university name, and marital status.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang W, Duan Y, Wang Y, Lippke S, Shang B, Lin Z, Wulff H, Baker JS. Psychosocial Mediators of Web-Based Interventions for Promoting a Healthy Lifestyle Among Chinese College Students: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2022 Sep 7;24(9):e37563. doi: 10.2196/37563. PMID 36069840
- [Derived] Duan Y, Liang W, Wang Y, Lippke S, Lin Z, Shang B, Baker JS. The Effectiveness of Sequentially Delivered Web-Based Interventions on Promoting Physical Activity and Fruit-Vegetable Consumption Among Chinese College Students: Mixed Methods Study. J Med Internet Res. 2022 Jan 26;24(1):e30566. doi: 10.2196/30566. PMID 35080497
- [Derived] Liang W, Duan YP, Shang BR, Wang YP, Hu C, Lippke S. A web-based lifestyle intervention program for Chinese college students: study protocol and baseline characteristics of a randomized placebo-controlled trial. BMC Public Health. 2019 Aug 13;19(1):1097. doi: 10.1186/s12889-019-7438-1. PMID 31409381

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03627949/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03627949/ICF_001.pdf